CLINICAL TRIAL: NCT01354795
Title: Prospective Study Comparing Methods of Obtainment of Specimen After EUS-FNA in Patients With Peri-pancreatic Mass
Acronym: EUS-FNA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Kwang Hyuck Lee / Department of Medicine, Dvision of Gastroenterology, Samsung Medical Center
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2010-07-219
Record Dates: First submitted 2011-04-24; First posted 2011-05-17 (Estimated); Last update posted 2011-05-17 (Estimated); Status verified 2011-05

CONDITIONS: Pancreatic Neoplasm; Neoplasm of Intra-abdominal Lymph Nodes
Keywords: EUS FNA; stylet; suction
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Suction; Endoscopic Ultrasound-Guided Fine Needle Aspiration

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1.EUS-FNA with or without suction (Experimental): During EUS FNA is performed, with or without self-retracting 10-mL syringe
  Interventions: Procedure: 1.EUS-FNA with or without suction
- 2.Pushing the stylet or injecting air (Experimental): EUS-FNA specimen is expelled from a needle with pushing the stylet into the needle or injecting air
  Interventions: Procedure: 2.Pushing the stylet or injecting air

INTERVENTIONS:
Procedure: 1.EUS-FNA with or without suction — During EUS-FNA of the peri-pancreatic mass was performed, with or without self-retracting 10-mL syringe applied.
  Other Names: EUS-FNA with or without suction
  Arms: 1.EUS-FNA with or without suction
Procedure: 2.Pushing the stylet or injecting air — EUS-FNA specimen is expelled from a needle with pushing the stylet or injecting air into the needle
  Other Names: Pushing the stylet or injecting air
  Arms: 2.Pushing the stylet or injecting air

SUMMARY:
EUS-guided FNA has been proved to be a safe and useful method for tissue sampling of gastrointestinal track lesions and other organ lesions including mediastinal and intra-abdominal lymph nodes, pancreas and hepatobiliary tree. The usefulness of EUS-FNA depends on several factors. For example, experience of the endosonographers, adequate sampling, sample preparing, accurate interpretation by the cytopathologist and on-site cytopathology interpretation. However, in many hospitals, no cytopathologist can be present during EUS-FNA. Therefore, determining appropriate methods to obtain and prepare EUS-guided FNA are important to make correct a diagnosis without on-site cytopathologist.

Suction with a self-retracting 10-mL syringe will likely bring in more cellularity but also more blood. Some endosonographers use no suction, others use constant suction. Usually specimen is expelled from a needle with pushing the stylet into the needle. But use of the stylet during EUS-FNA is difficult and time consuming process. Injecting air was not recommended, because of spraying out uncontrollably, increasing risk of air artifact and specimen clotting. However, there is no further study which one is the appropriate, suction or no suction and pushing the stylet or injecting air until now.

The hypothesis and aim of the prospective randomized controlled trials are as follows:

First hypothesis: There was no difference in the adequacy, cellularity, bloodiness, contamination, air artifact in specimen obtained by each methods, suction or no suction and pushing the stylet or injecting air.

Aim #1 : To compare the adequacy, cellularity, bloodiness, contamination, air artifact in specimen obtained by each methods, suction or no suction and pushing the stylet or injecting air.

Second hypothesis: There was no difference in sensitivity, specificity, diagnostic accuracy, positive predictive value, negative predictive value and statistical agreement in specimen obtained by each methods, suction or no suction and pushing the stylet or injecting air.

Aim #2 : To compare the sensitivity, specificity, diagnostic accuracy, positive predictive value, negative predictive value and statistical agreement in specimen obtained by each methods, suction or no suction and pushing the stylet or injecting air.

DETAILED DESCRIPTION:
On-site cytopathology interpretation during EUS-FNA has a significant clinical impact by increasing the diagnostic yield of the FNA. However, many hospitals do not have provision for on- site diagnosis of EUS FNA specimen. Therefore, optimal specimen obtainment and preparation of EUS FNA are is important to accurate diagnosis. EUS FNA is performed with or without self-retracting 10-mL syringe according to endosonographer's preference. In general, if there is too little cellularity on immediate cytologic evaluation, then use more suction, and, conversely, if the samples are too bloody, then use less suction. However, it is hard to determine the quality of specimen without on-site cytopathology interpretation. The actual way material is expressed from the needle may influence yield. Injecting air to express the material is problematic, because the material may spray out uncontrollably, risk of air artifact and specimen clotting may increase . A more controlled method is to pushing the stylet and slowly advance it to the needle tip. But use of the stylet during EUS-FNA is not only difficult and time consuming process but also increasing the risk of accidental needle stick injury. However, there is no firm evidence which one is the appropriate, suction or no suction and pushing the stylet or injecting air. If there was no significant difference between each methods, appropriate methods of obtaining and preparing aspirates undergoing EUS-FNA is no suction and injecting air and EUS FNA may perform more easier and shorter.

In this prospective randomized controlled trial, patients with peripancreatic mass for EUS-FNA will be included. One patient will be underwent at least four puncture during EUS-FNA. The sequence of EUS-FNA with first four methods will be selected by using a randomization scheme obtained from a sealed envelope : (1) negative pressure suction with 10 mL syringe and pushing the stylet; (2) negative pressure suction with 10 mL syringe and injecting air; (3) without negative pressure suction and pushing the stylet; (4) without negative pressure suction and injecting air. EUS FNA will be performed by two experienced endosonographers. All specimens will be read by same experienced pathologist blinded to methods.

The investigators will compare between the four groups in terms of adequacy, cellularity, bloodiness, contamination, air artifact. The sensitivity, specificity, diagnostic accuracy, positive predictive value, negative predictive value and statistical agreement for the different methods will be calculated.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than 18 years
2. Presence of peri pancreatic mass, mediastinal or intra-abdominal lymphadenopathy confirmed by investigational modality - CT scan, magnetic resonance imaging, EUS.
3. Capable of providing informed consent

Exclusion Criteria:

1. Severe coagulopathy (INR > 1.5) or thrombocytopenia (platelet count < 50,000)
2. History of acute pancreatitis in the preceding 4 weeks
3. Pregnancy
4. Inability to provide informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2010-09; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Compare the degree of cytologic quality in specimen obtained by EUS-FNA with or without suction, pushing the stylet or injecting air. | within 6 months
  The primary endpoint of this study is to determine that there is no difference in cytologic quality of FNA specimens with or without suction, pushing the stylet or injecting air: to compare the adequacy, cellularity, bloodiness, contamination, air artifact in specimen obtained by each methods.

SECONDARY OUTCOMES:
Compare the diagnostic yield in specimen obtained by EUS-FNA with or without suction, pushing the stylet or injecting air. | within 6 months
  The secondary endpoint of this study is to determine that there is no difference in diagnostic yield of FNA specimens with or without suction, pushing the stylet or injecting air: to compare the sensitivity, specificity, diagnostic accuracy, positive predictive value, negative predictive value and statistical agreement in specimen obtained by each methods.

CONTACTS AND LOCATIONS:
Overall Officials: Kwang Hyuck Lee, M.D., Study Director — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Lee JK, Choi JH, Lee KH, Kim KM, Shin JU, Lee JK, Lee KT, Jang KT. A prospective, comparative trial to optimize sampling techniques in EUS-guided FNA of solid pancreatic masses. Gastrointest Endosc. 2013 May;77(5):745-51. doi: 10.1016/j.gie.2012.12.009. Epub 2013 Feb 21. PMID 23433878